CLINICAL TRIAL: NCT04311840
Title: Impact of Nimodipine on Sublingual Microcirculation in Patients With Subarachnoid Hemorrhage - a Prospective Monocentric Observational Study
Brief Title: Impact of Nimodipine on Sublingual Microcirculation in Patients With Hemorrhage - a Prospective Monocentric Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Sponsor
Other Study IDs: SAH_Nimodipine
Record Dates: First submitted 2019-11-18; First posted 2020-03-17 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Subarachnoid Hemorrhage
Keywords: nimodipine; sublingual microcirculation; Side-stream Dark Field imaging
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SAH patients with nimodipine: Patients with SAH receiving nimodipine as prevention of vasospasms and as a nootropic drug.
- SAH patients without nimodipine: Patients with SAH not receiving nimodipine as prevention of vasospasms and as a nootropic drug or in whom the drug has been temporarily discontinued.

SUMMARY:
Nimodipine can increase Functional Capillary Density (FCD) as a parameter of the sublingual microcirculation in patients with subarachnoid hemorrhage (SAH) compared to patients without nimodipine.

DETAILED DESCRIPTION:
SAH group - in patients with SAH and documented vasospasms by digital subtraction angiography (DSA) of trans-cranial doppler imaging (TCD) of arteria cerebri media nimodipine is indicated because it is proven to improve the clinical outcome. The disfunction of cerebral microcirculation in rats with SAH has been documented [1-6]. Changes in sublingual microcirculation in patients with SAH with documented vasospasms with nimodipine has not been described.

ELIGIBILITY:
Inclusion Criteria:

* adulthood
* ICU admission
* diagnosis of non-traumatic subarachnoid hemorrhage

Exclusion Criteria:

* inherited coagulation disorder
* rheumatic disease
* microangiopathy
* patient of representative refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted to the neurosurgical ICU with the diagnosis of subarachnoid hemorrhage. Might be alert, somnolent or sedated on mechanical ventilation. Might be after endovascular coiling or surgical clipping of the aneurysm.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional capillary density (FCD) | One week
  Parameter describing the perfusion of the microcirculation
Proportion of perfused vessels (PPV) | One week
  Parameter describing the perfusion of the microcirculation

SECONDARY OUTCOMES:
Vasospasm occurence | One week
  Occurence of vasospasms on angiography and/or transcranial Doppler
Circulatory incoherence | One week
  Deranged microcirculation in patients on catecholamines

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Třebeš, Czechia

IPD SHARING:
Plan to Share IPD: No